CLINICAL TRIAL: NCT06538883
Title: Efficacy and Safety of Ciprofol Versus Propofol for Sedation in ICU Patients With Mechanical Ventilation: A Multi-Center, Double-Blind, Randomized Controlled Trial
Brief Title: Sedation in ICU Patients With Mechanical Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Collaborators: The First Affiliated Hospital of Air Force Medicial University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Zhongnan University Xiangya Second Hospital (Unknown); Renmin Hospital of Wuhan University (Other); First Affiliated Hospital of Suzhou Medical College (Other); The First Affiliated Hospital of Nanchang University (Other); The Third Bethune Hospital of Jilin University (Unknown); Zhongnan Hospital (Other); First Affiliated Hospital of the University of Science and Technology of China (Anhui Provincial Hospital) (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Kunming Medical University (Other); Sichuan Academy of Medical Sciences (Other); Anhui provincial chest hospital (Unknown); The Guangxi Zhuang Autonomous Region People's Hospital (Unknown); Second Affiliated Hospital of Suzhou University (Other); The Ninth People's Hospital of Suzhou (Unknown); Fifth Affiliated Hospital of Xinjiang Medical University (Other); Xuzhou Medical University Hospital (Unknown); First People's Hospital of Hangzhou (Other); Hebei Medical University Fourth Hospital (Other); Huai'an First People's Hospital (Other); Jinan City People's Hospital (Unknown); The First People's Hospital of Lianyungang (Other); Jiangsu Subei People's Hospital (Unknown); Suqian First Hospital (Other); Tai'an City Central Hospital (Unknown); Xuzhou Central Hospital (Other); The first People's Hospital of Yancheng City (Unknown); The First People's Hospital of Zunyi (Other); Jiangxi Provincial People's Hopital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Fei Peng, Principal Investigator, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAME study
Record Dates: First submitted 2024-07-04; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Respiration, Artificial; Hypnotics and Sedatives
Keywords: Sedation; Mechanical Ventilation; ICU; Ciprofol; Propofol
MeSH Terms: conditions — Respiratory Aspiration | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol (Experimental)
  Interventions: Drug: Sedation with Ciprofol
- Propofol (Active Comparator)
  Interventions: Drug: Sedation with Propofol

INTERVENTIONS:
Drug: Sedation with Ciprofol — During the drug administration period, ciprofol were IV infused at loading doses of 0.1 mg/kg, respectively, over 4 minutes ± 30 seconds depending on the physical condition of each patient. Ciprofol were then immediately administered at an initial maintenance dose of 0.3 mg/kg/hr, with a target sedation depth of RASS +1 to -2, based on the Pain, Agitation/sedation, Delirium, Immobility (rehabilitation/mobilization), and Sleep (disruption) guideline.
  Arms: Ciprofol
Drug: Sedation with Propofol — During the drug administration period, propofol were IV infused at loading doses of 0.5 mg/kg, respectively, over 4 minutes ± 30 seconds depending on the physical condition of each patient. Propofol were then immediately administered at an initial maintenance dose of 1.5 mg/kg/hr, with a target sedation depth of RASS +1 to -2, based on the Pain, Agitation/sedation, Delirium, Immobility (rehabilitation/mobilization), and Sleep (disruption) guideline.
  Arms: Propofol

SUMMARY:
Sedatives are the mostly common prescription for patients with mechanical ventilation due to the disease or therapies.

Ciprofol is a new intravenous anesthetic agent transformed from propofol, and has a similar sedative effect of propofol in previous study.

Whether ciprofol is safe and effective similar with propofol for sedation in ICU patients with mechanical ventilation? Therefor, a multi-center, double-blind, randomized control trial was conducted with a noninferiority design, to compared the rate of successful sedation without hypotension of sedation by ciprofol or propofol in ICU patients with mechanical ventilation.

A Multi-Center, Double-Blind, Randomized Controlled Trial will be launched to evaluate the efficacy and safety of ciprofol versus propofol for sedation in ICU patients with mechanical ventilation.

ELIGIBILITY:
Inclusion criteria (patients who met all the following criteria):

1. Adults are sequentially admitted to ICU undergoing mechanical ventilation; Patients are expected to need 6-24 hours of sedation for the target RASS ranged from +1 to -2 after randomization;
2. Aged ≥ 18 and ≤ 80 years old, with no gender requirement;
3. The patients or their family members fully understood the objectives and significance of this study and voluntarily participated and signed informed consent forms.

Exclusion criteria (patients who met 1 of the following criteria were excluded):

1. Patients known to be allergic or contraindicated to ciprofol. 2. BMI<18 kg/m2 or >30 kg/m2. 3. Patients who had received sedation for more than 3 days in an ICU or in a general ward prior to being transferred to the ICU before signing an informed consent form.

4. Patients have the following medical history or evidence of any of the following conditions at screening, which may increase the sedation/anesthesia risk:

1. Cardiovascular system: New York Heart Association (NYHA) Class III and IV heart failure, Adams-stokes syndrome; patients who required vasopressor (equivalent norepinephrine ≥ 1μg/kg/min) to maintain a normal blood pressure.
2. Patients with hepatic and renal failure (liver function: refer to Child-Pugh grade C; renal function: eGFR ≤ 30 mL/(min·1.73 m2) [eGFR was calculated using the Modification of Diet in Renal Disease (MDRD) equation: eGFR = 175 × serum creatinine (SCr) - 1.234 × age - 0.179 × 0.79 (females)]; patients undergoing dialysis.
3. Patients with grand mal epilepsy and convulsion; a Glasgow coma scale (GCS) ≤ 12 points.

5. Patients with an expected survival of ≤ 24 h. 6. Pregnant or lactating females. 7. Patients participated in other drug clinical trials before screening. 8. Other conditions that patients were judged by the investigator to be unsuitable for inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the rate of successful sedation without hypotension | within the first 30 minutes of administering the study drug
  The primary outcome is the rate of successful sedation without hypotension, which have to meet the following three criteria simultaneously: 1) Sedation within the RASS target (+1 to -2); 2) No rescue therapy is used; 3) No hypotension occurs, within the first 30 minutes of administering the study drug.

SECONDARY OUTCOMES:
the rate of within sedation target (RASS: +1 to -2) without hypotension in the first 1hour of administering the study drug; | within the first 1hour of administering the study drug
the rate of within sedation target (RASS: +1 to -2) without circulatory inhibition (defined as either hypotension or bradycardia) in the first 1hour of administering the study drug; | within the first 1hour of administering the study drug
Usage of study drugs | within the first 24hours of administering the study drug
  the total additional dose will be recorded;
Duration of mechanical ventilation | from intubation (for patients intubated after ICU admission) or ICU admission (for patients admitted with intubation) until the date of first estubation or date of death from any cause, whichever came first, assessed up to 28 days
  Duration of mechanical ventilation: defined as the time from intubation (for patients intubated after ICU admission) or ICU admission (for patients admitted with intubation) to extubation;
Extubation time | from intubation (for patients intubated after ICU admission) or ICU admission (for patients admitted with intubation) to extubation
  time from stopping the study drug to extubation; not applicable for patients who withdraw early or do not plan to extubate after stopping the drug;
Awakening time | from stopping the study drug until the time of awakening from sedation (RASS ≥ 0) or death from any cause, whichever came first, assessed up to 28 days
  defined as the time from stopping the study drug to awakening from sedation (RASS ≥ 0). If RASS is ≥ 0 at the time of stopping the drug, the awakening time is recorded as 0;
Incidence of delirium | from administation of study drug until the time of awakening from sedation (RASS ≥ 0) or death from any cause, whichever came first, assessed up to 28 days
  Incidence of delirium, which is assessed using the CAM-ICU;
Length of ICU stay | the time from ICU admission to discharge from the ICU or death from any cause, whichever came first, assessed up to 28 days
  defined as the time from ICU admission to discharge from the ICU;
The 28-day mortality | from administation of study drug to 28 days
  all caused mortality within 28 days.
Incidence of hypotension | from the time of signing informed consent to 2 hours after the end of study drug administration
  Hypotension was defined as SBP < 90 mmHg, or DBP < 60 mmHg, or MAP < 70 mmHg, or a drop of more than 30% from baseline, more than 2 minutes, or as determined by the investigator; and the use of vasopressor medications will be recorded;
Incidence of bradycardia | from the time of signing informed consent to 2 hours after the end of study drug administration
  HR < 40 bpm or a drop of more than 30% from baseline; the use of medications for bradycardia intervention

IPD SHARING:
Plan to Share IPD: Undecided